CLINICAL TRIAL: NCT04150445
Title: Internet Treatment for Overweight and Obese Patients - a Pilot Study
Brief Title: Internet Treatment for Persons With Overweight or Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 272763
Record Dates: First submitted 2019-10-23; First posted 2019-11-04 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Body Weight
MeSH Terms: conditions — Overweight; Obesity; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet treatment for overweight and obese patients (Experimental): The intervention is a treatment of overweight and obesity based on cognitive behavioural therapy provided via the Internet. The treatment lasts for six months and comprises 12 treatment modules. The patient works with each module for two weeks. The modules conclude with one or more exercise tasks to be performed before the next module is activated. The patient has written contact with the therapist via the Internet platform.
  Interventions: Behavioral: Internet treatment for overweight and obese patients

INTERVENTIONS:
Behavioral: Internet treatment for overweight and obese patients — The behavioral treatment is provided via the Internet and comprises 12 modules that the patient follows for 6 months. The treatment modules include self-monitoring, goal setting, relapse prevention, psycho-education about nutrition, eating behavior, physical activity, sleep and stress management. Each module ends with one or more exercises to be completed before the next module is activated.

SUMMARY:
Overweight and obesity are increasing and more than 50% of all people over 18 years in Sweden are overweight or obese. Main causes are changes in lifestyle habits regarding diet and physical activity. Obesity increases the risk of various diseases such as type 2 diabetes, cardiovascular disease, arthrosis and cancer; it also affects the quality of life. Losing 5-10% of body weight can improve metabolic health and quality of life. However, weight loss is difficult to achieve and especially to maintain over a longer period of time. Treatment based on cognitive behavioral therapy improves long-term outcomes. A behavioral treatment program via the Internet has been developed that contains 12 treatment modules that the patient follows for 6 months. The patient has regular contact with a therapist who follows the patient's treatment process and provides support. The purpose of this pilot study is to evaluate the Internet-based treatment regarding weight reduction, change in eating habits, physical activity and quality of life. We also intend to investigate how feasible and user-friendly the treatment program is and the patients' experiences of the treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* BMI 30 or over
* BMI over 28 and under 30 with one or more of the following: hypertension, prediabetes, type 2 diabetes, coronary heart disease, hyperlipidaemia, liver steatosis, sleep apnea or polycystic ovary syndrome

Exclusion Criteria:

* Severe mental illness
* Previous or present eating disorder
* Pregnancy
* Breast feeding
* Serious cancer under treatment
* Use of weight-loss drugs
* Weight loss treatment in the last 6 months
* Misuse of alcohol or drugs
* Type 1 diabetes
* Not being able to speak/read/write Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Body weight | Change from baseline to follow-up at 6 months and 12 months
  Weight reduction in kg

SECONDARY OUTCOMES:
Dietary habits | Change from baseline to follow-up at 6 months and 12 months
  Change in dietary habits measured by a questionnaire from the National Board of Health and Welfare, Sweden. The questionnaire includes five questions about how often the person eats vegetables, fruits, fish, sweets and breakfast.
Physical activity | Change from baseline to follow-up at 6 months and 12 months
  Change in physical activity measured with a questionnaire from The National Board of Health and Welfare, Sweden. The questionnaire contains two questions about exercise and everyday activities that measure how much time per week the person performs: 1) strenuous activities, e.g. running, playing ball, and 2) moderately strenuous activities, e.g. walking, cycling.
Psychosocial functioning | Change from baseline to follow-up at 6 months and 12 months
  Change in weight-related psychosocial functioning measured by the Obesity-related Problems scale, version 3 (OPv3). OPv3 comprises 26 items on a four-point response scale. The participants indicate how bothered they are by their obesity in a broad range of social activities and to what extent they avoid social activities because of their obesity. The responses are aggregated into two domains: Distress (13 items) and Avoidance (13 items). Scale scores range from 0 (no distress/avoidance) to 100 (maximum distress/avoidance).
Experiences of the treatment program | From treatment start to follow-up after treatment ends at 6 months
  The patient's experiences of the treatment program are measured with five study-specific questions about how easy or difficult it was 1) to follow the treatment program, 2) to understand the language and content, 3) to use the program 4) to understand the home tasks and if they were relevant, and 5) how useful feedback from the therapist was .
Experiences of the treatment effects | From baseline to follow-up at 6 months and 12 months
  The patient's experiences of the treatment effects are measured with study-specific questions (18 and 15 questions at 6 and 12 months follow-up respectively). The questions concern the following aspects: 1) if the treatment has been helpful in making lifestyle changes, 2) if the participant is satisfied or dissatisfied with the weight change, 3) if the participant considers that the treatment has had an effect on health and well-being.

OTHER OUTCOMES:
Causes of drop-out from treatment | Within two weeks of the end of treatment
  Interviews with participants who finish the treatment prematurely

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Jansson, MD, PhD, Principal Investigator — Region Örebro County
Locations (1):
- Obesity Unit, Örebro University Hospital, Region Örebro County, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No